CLINICAL TRIAL: NCT00705575
Title: A 12 Week, Double-blind, Randomized, Parallel Group, Multi-center Study to Evaluate the Efficacy and Safety of the Combination of Aliskiren 300 mg and Hydrochlorothiazide 25 mg Compared to Aliskiren 300 mg in Patients With Stage II Hypertension
Brief Title: Efficacy and Safety of the Combination Aliskiren (300 mg) and Hydrochlorothiazide (25mg) to Aliskiren (300mg) Monotherapy in Patients With Staged II Hypertension
Acronym: ACQUIRE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Novartis, Novartis
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CSPP100A2353
Record Dates: First submitted 2008-06-23; First posted 2008-06-26 (Estimated); Results first posted 2011-01-21 (Estimated); Last update posted 2011-05-30 (Estimated); Status verified 2011-05

CONDITIONS: Hypertension
Keywords: Essential Hypertension; Stage II
MeSH Terms: conditions — Hypertension; Essential Hypertension | interventions — aliskiren; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aliskiren/hydrochlorothiazide (HCTZ) (300/25 mg) (Experimental)
  Interventions: Drug: Aliskiren/hydrochlorothiazide (HCTZ) (300/25 mg)
- Aliskiren (300 mg) (Active Comparator)
  Interventions: Drug: Aliskiren (300 mg)

INTERVENTIONS:
Drug: Aliskiren/hydrochlorothiazide (HCTZ) (300/25 mg) — During the titration period, patients received aliskiren/hydrochlorothiazide (HCTZ) 150/12.5 mg for 1 week.
  Arms: Aliskiren/hydrochlorothiazide (HCTZ) (300/25 mg)
Drug: Aliskiren (300 mg) — During the titration period, patients received aliskiren 150 mg for one week. Subsequently, patients were up-titrated and received aliskiren 300 mg.
  Arms: Aliskiren (300 mg)

SUMMARY:
This study will compare the efficacy and safety of once daily dosing of aliskiren monotherapy to once daily dosing of aliskiren and hydrochlorothiazide combination therapy in patients with Stage II hypertension over a period of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients ≥18 years of age.
* Patients with a diagnosis of Stage II hypertension, defined as mean sitting Systolic Blood Pressure (msSBP) ≥ 160 mmHg and < 180 mmHg at Visit 2.

Exclusion Criteria:

* Severe hypertension defined as msSBP ≥ 180 mmHg and/or mean sitting Diastolic Blood Pressure (msDBP) ≥ 110 mmHg.
* Secondary form of hypertension.
* Current diagnosis of heart failure (New York Heart Association [NYHA] Class II-IV).
* Current angina pectoris requiring pharmacological therapy (other than stable doses of oral or topical nitrates).
* Second or third degree heart block without a pacemaker.
* Concurrent potentially life threatening arrhythmia or symptomatic arrhythmia, atrial fibrillation or atrial flutter, during the 12 months prior to Visit 1.
* Clinically significant valvular heart disease.
* Previous history of hypertensive encephalopathy or stroke, Transcient Ischemic Attack (TIA), heart attack, coronary bypass surgery or any PCI.
* Known Keith-Wagener grade III or IV hypertensive retinopathy.
* In the month prior to Visit 1, patients on combination antihypertensive therapy that includes more than 2 classes of antihypertensive medications.
* Patients on combined antihypertensive medication that contain two classes of antihypertensive medications are considered to take two antihypertensive medications.
* Inability to discontinue prior antihypertensive or other CV medications as required by the protocol.
* Patients with Type 1 diabetes mellitus.
* Patients with Type 2 diabetes mellitus not well controlled .
* Elevated Serum potassium (over 5.3 mEq/L (mmol/L).
* Any surgical or medical condition or the use of any medication which might significantly alter the absorption, distribution, metabolism, or excretion of study drugs.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 688 (Actual)
Dates: Start 2008-06; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- Investigative Site, East Hanover, New Jersey, United States
- Investigative Site, Buenos Aires, Argentina
- Investigative Site, Quito, Ecuador
- Investigative Site, Berlin, Germany
- Investigative Site, Guatemala City, Guatemala
- Investigative Site, Rome, Italy
- Investigative Site, Basel, Switzerland
- Investigative Site, Ankara, Turkey (Türkiye)

RESULTS

PARTICIPANT FLOW:
Groups:
- Aliskiren/Hydrochlorothiazide (HCTZ) (300/25 mg): During the titration period, patients received aliskiren/hydrochlorothiazide (HCTZ) 150/12.5 mg for 1 week. Subsequently, patients were up-titrated and received aliskiren/HCTZ 300/25 mg.
Period: Overall Study
Arm/Group | Aliskiren/Hydrochlorothiazide (HCTZ) (300/25 mg) | Aliskiren (300 mg)
Started | 349 | 339
Completed | 326 | 293
Not Completed | 23 | 46
Not completed — Abnormal laboratory value(s) | 0 | 3
Not completed — Abnormal test procedure result(s) | 2 | 12
Not completed — Adverse Event | 11 | 15
Not completed — Lost to Follow-up | 3 | 4
Not completed — Protocol Violation | 2 | 2
Not completed — Withdrawal by Subject | 5 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aliskiren/Hydrochlorothiazide (HCTZ) (300/25 mg) | Aliskiren (300 mg) | Total
Number analyzed (Participants) | 349 | 339 | 688
Age Continuous [Mean (Standard Deviation); unit: years] | 57.4 (10.33) | 56.4 (10.73) | 56.9 (10.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 169 | 172 | 341
  Male | 180 | 167 | 347

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Sitting Systolic Blood Pressure (msSBP) From Baseline to End of Study (Week 12)
Description: At the first visit, blood pressure (BP) was measured in both arms and the arm having the higher BP reading was the arm used for all subsequent readings throughout the study. Patients were required to sit for five minutes with feet flat on the floor, with arm resting so that the bottom of the cuff was at the same level as the heart. BP was measured three times at 1 to 2-minute intervals at each visit using the correct cuff size. The mean BP was calculated from the 3 readings.
Time Frame: Baseline to end of study (Week 12)
Population: Full analysis set (FAS): All randomized patients. For each patient, the last post-baseline measurement during the double-blind period was carried forward. n = number of patients with non-missing Week 12 measurement or last observation carried forward (LOCF) value.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Aliskiren/Hydrochlorothiazide (HCTZ) (300/25 mg) | Aliskiren (300 mg)
Number analyzed (Participants) | 346 | 335
mm Hg | -30.01 (1.053) | -20.29 (1.067)

2. Secondary Outcome: Change in Mean Sitting Systolic Blood Pressure (msSBP) From Baseline to Week 8
Description: as for outcome 1
Time Frame: Baseline to Week 8
Population: Full analysis set (FAS): All randomized patients. For each patient, the last post-baseline measurement during the double-blind period was carried forward. n = number of patients with non-missing Week 8 measurement or last observation carried forward (LOCF) value.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Aliskiren/Hydrochlorothiazide (HCTZ) (300/25 mg) | Aliskiren (300 mg)
Number analyzed (Participants) | 346 | 335
mm Hg | -30.09 (1.079) | -20.75 (1.094)

3. Secondary Outcome: Change in Mean Sitting Diastolic Blood Pressure (msDBP) From Baseline to Week 8 and to Week 12
Description: as for outcome 1
Time Frame: Baseline to Week 12
Population: Full analysis set (FAS): All randomized patients. For each patient, the last post-baseline measurement during the double-blind period was carried forward. n = number of patients with non-missing Week 8 or Week 12 measurement or last observation carried forward (LOCF) value.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Aliskiren/Hydrochlorothiazide (HCTZ) (300/25 mg) | Aliskiren (300 mg)
Number analyzed (Participants) | 346 | 335
mm Hg
  Baseline to Week 8 | -13.69 (0.599) | -7.99 (0.607)
  Baseline to Week 12 | -12.64 (0.590) | -8.18 (0.598)

4. Secondary Outcome: Percentage of Patients Achieving the Target Blood Pressure (msSBP < 140 mm Hg and msDBP < 90 mm Hg, and msSBP < 130 mm Hg and msDBP < 80 mm Hg for Diabetics) at Week 8 and Week 12
Description: as for outcome 1
Time Frame: Baseline to Week 12
Population: as for outcome 3
Measure: Number; unit: Percentage
Arm/Group | Aliskiren/Hydrochlorothiazide (HCTZ) (300/25 mg) | Aliskiren (300 mg)
Number analyzed (Participants) | 346 | 335
Percentage
  Baseline to Week 8 | 53.5 | 30.4
  Baseline to Week 12 | 54.6 | 32.2

ADVERSE EVENTS:
Arm/Group | Aliskiren/Hydrochlorothiazide (HCTZ) (300/25 mg) | Aliskiren (300 mg)
Serious Adverse Events (participants affected / at risk) | 2/349 | 4/339
Other Adverse Events (participants affected / at risk) | 27/349 | 34/339
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren/Hydrochlorothiazide (HCTZ) (300/25 mg) (N=349) | Aliskiren (300 mg) (N=339)
Vertigo (Ear and labyrinth disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Fracture displacement (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren/Hydrochlorothiazide (HCTZ) (300/25 mg) (N=349) | Aliskiren (300 mg) (N=339)
Dizziness (Nervous system disorders) | 19 | 10
Headache (Nervous system disorders) | 14 | 29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.